CLINICAL TRIAL: NCT04051450
Title: Immune Checkpoints in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHEUNG, Siu Tim, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: CRC_immune2018
Record Dates: First submitted 2019-07-28; First posted 2019-08-09 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood sample (10ml peripheral blood) will be drawn before the operation or endoscopic session. A small portion of the tumor and non-tumor tissue tissues from resected specimens or biopsy tissues will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) ranked the first in cancer incidence in Hong Kong and it is frequently lethal with heterogeneous drug responses and survival outcomes. Immune-based approaches targeting to enhance tumor-specific responses have been actively under investigation as therapeutic strategies. Currently, PD1 and PD-L1 blockade has shown promising results in clinical trials especially in colorectal cancer patients with microsatellite instability. This study aims to examine the role of PD-L1/PD1 in immune cell-mediated cytotoxicity in colorectal cancer patients.

DETAILED DESCRIPTION:
Aim: To examine the role of PD-L1/PD1 in immune cell-mediated cytotoxicity in colorectal cancer patients.

Objectives: 1. Comprehensive investigation of PD-L1/PD1 in colorectal cancer in association with chemotherapy responses and immune activities; 2. Examine the functional role of PD-L1/PD1 targeting in immune cell-mediated cytotoxicity.

Hypothesis: It is hypothesized that PD-L1/PD1 has pivotal role on the immune cell-mediated cytotoxicity in colorectal cancer.

Significances: The current study will elucidate the significance of PD-L1/PD1 on chemo-resistance and the effect on immune cells and their functional properties. The study will enhance the understanding on chemotherapy response and immune evasion. The long-term goal is to provide the crucial information on oncoimmunology to improve efficacy of immunotherapy in cancer treatment.

Subjects: Only those patients for whom colorectal cancer is the indicated clinical diagnosis will be recruited in the current study. Possible participants will be patients undergoing tumor resection or endoscopic examination at the Department of Surgery, Prince of Wales Hospital, Shatin, Hong Kong. Specimens will be collected from sixty-eight colorectal cancer patients. The estimated duration for collection of all the necessary samples will be two years. With at least one year of follow-up information, the proposed study should be completed in three years. For the current study, single blood sample (10 ml of peripheral blood in EDTA) will be drawn before the operation or endoscopic session. A small portion of the tumor and non-tumor tissue tissues from resected specimens or biopsy tissues will be collected for histological evaluation, primary culture and for comparison of the genetic and protein components in the blood specimen.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer patients undergoing resection or endoscopic examination at the Department of Surgery, Prince of Wales Hospital, Shatin, Hong Kong

Exclusion Criteria:

* patients who do not consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients undergoing resection or endoscopic examination at the Department of Surgery, Prince of Wales Hospital, Shatin, Hong Kong
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Generation of candidate biomarkers PD-L1/PD1/GEP by laboratory assay qPCR for prognostication. | Three years.
  Biomarkers PD-L1/PD1/GEP will be investigated by laboratory assay real-time quantitative PCR. The biomarker levels in tissue specimens and the association with recurrence-free survival will be analyzed for prognostication.

CONTACTS AND LOCATIONS:
Overall Officials: ST Cheung, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Farkona S, Diamandis EP, Blasutig IM. Cancer immunotherapy: the beginning of the end of cancer? BMC Med. 2016 May 5;14:73. doi: 10.1186/s12916-016-0623-5. PMID 27151159
- [Background] Passardi A, Canale M, Valgiusti M, Ulivi P. Immune Checkpoints as a Target for Colorectal Cancer Treatment. Int J Mol Sci. 2017 Jun 21;18(6):1324. doi: 10.3390/ijms18061324. PMID 28635639
- [Background] Brenner H, Kloor M, Pox CP. Colorectal cancer. Lancet. 2014 Apr 26;383(9927):1490-1502. doi: 10.1016/S0140-6736(13)61649-9. Epub 2013 Nov 11. PMID 24225001
- [Background] Guinney J, Dienstmann R, Wang X, de Reynies A, Schlicker A, Soneson C, Marisa L, Roepman P, Nyamundanda G, Angelino P, Bot BM, Morris JS, Simon IM, Gerster S, Fessler E, De Sousa E Melo F, Missiaglia E, Ramay H, Barras D, Homicsko K, Maru D, Manyam GC, Broom B, Boige V, Perez-Villamil B, Laderas T, Salazar R, Gray JW, Hanahan D, Tabernero J, Bernards R, Friend SH, Laurent-Puig P, Medema JP, Sadanandam A, Wessels L, Delorenzi M, Kopetz S, Vermeulen L, Tejpar S. The consensus molecular subtypes of colorectal cancer. Nat Med. 2015 Nov;21(11):1350-6. doi: 10.1038/nm.3967. Epub 2015 Oct 12. PMID 26457759
- [Background] Llosa NJ, Cruise M, Tam A, Wicks EC, Hechenbleikner EM, Taube JM, Blosser RL, Fan H, Wang H, Luber BS, Zhang M, Papadopoulos N, Kinzler KW, Vogelstein B, Sears CL, Anders RA, Pardoll DM, Housseau F. The vigorous immune microenvironment of microsatellite instable colon cancer is balanced by multiple counter-inhibitory checkpoints. Cancer Discov. 2015 Jan;5(1):43-51. doi: 10.1158/2159-8290.CD-14-0863. Epub 2014 Oct 30. PMID 25358689